CLINICAL TRIAL: NCT02621541
Title: Dual Tracer Functional Imaging of Nonfunctional Pancreatic Neuroendocrine Tumors Using 68Ga-DOTA-NOC and 18F-FDG PET/CT
Brief Title: Nonfunctional Pancreatic NET and PET Imaging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P-NETPET
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Diagnosis
Keywords: neuroendocrine tumor; pancreas; diagnosis; positron emission tomography
MeSH Terms: conditions — Disease; Neuroendocrine Tumors | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preoperative diagnosis (Experimental): Preoperative diagnosis
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT

SUMMARY:
Predicting aggressive behavior in the group of nonfunctional pancreatic neuroendocrine tumors (NF P-NET) remains a difficult problem in clinical practice. At present, the treatment planning in P-NET is significantly restricted by the limited results of conventional imaging. In addition, increasing use of multidetector computed tomography (MDCT) and magnetic resonance imaging (MRI) is increasing the number of NF P-NETs detected. Somatostatin receptor scintigraphy (SRS) combined with anatomical imaging are the conventional modalities in imaging of P-NET, but by these methods the diagnostic accuracy still remains compromised. Furthermore, recently encouraging results have been obtained in P-NET using 68Ga-labelled somatostatin analog, DOTA-1-NaI3-octreotide (68Ga-DOTANOC) positron emission tomography-computed tomography (PET-CT).

The aim of the current project is to evaluate the possibility to enhance the diagnostic accuracy by using dual trace functional imaging 18F-labelled fluorodeoxyglucose (18F-FDG) and 68Ga-DOTANOC PET-CT imaging in patients with NF P-NET. The study consists of 20 patients with NF P-NET. The patients enrolled in the study will be imaged 68Ga-DOTANOC and 18F-FDG PET-CT followed by surgery or follow-up with endoscopic ultrasonography (EUS) biopsies. The data will be collected between autumn 2015 and spring 2018.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of nonfunctional P-NET on primary CT (i.e hypervascularity) or MRI
* signed informed consent

Exclusion Criteria:

* vulnerable study subjects such as described in Finnish law concerning clinical studies (disabled, children, pregnant or breast-feeding women, prisoners) will not be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The SUV of 68Ga-DOTANOC and 18F-FDG PET-CT predict the malignant potential of P-NETs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Saila Kauhanen, MD, PhD, Principal Investigator — Turku University Hospital
Locations (2):
- Finland (2):
  - Turku Division of Digestive Surgery and Urology, Turku, Turku
  - HUS Vatsakeskus, Helsinki

REFERENCES:
- [Derived] Majala S, Seppanen H, Kemppainen J, Sundstrom J, Schalin-Jantti C, Gullichsen R, Schildt J, Mustonen H, Vesterinen T, Arola J, Kauhanen S. Prediction of the aggressiveness of non-functional pancreatic neuroendocrine tumors based on the dual-tracer PET/CT. EJNMMI Res. 2019 Dec 23;9(1):116. doi: 10.1186/s13550-019-0585-7. PMID 31872324